CLINICAL TRIAL: NCT05583032
Title: A Randomised Prospective Evaluation of the Long-Term Impact of Assistive Artificial Intelligence on Anaesthetists' Ultrasound Scanning for Regional Anaesthesia
Brief Title: An Evaluation of the Long-Term Impact of Assistive AI on Anaesthetists' Ultrasound Scanning for UGRA
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2022_AG_10
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Ultrasound Imaging of Anatomical Structures
Keywords: ScanNav; Anatomy PNB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ScanNav Anatomy PNB aided: Participants completing scans for regional anaesthesia with the aid of ScanNav Anatomy PNB.
  Interventions: Device: ScanNav Anatomy PNB
- ScanNav Anatomy PNB unaided: Participants completing scans for regional anaesthesia without the aid of ScanNav Anatomy PNB.

INTERVENTIONS:
Device: ScanNav Anatomy PNB — AI-powered device that highlights anatomy of interest during ultrasound scans.
  Groups: ScanNav Anatomy PNB aided

SUMMARY:
A randomised, blinded interventional prospective study evaluating the long-term impact of assistive artificial intelligence on anaesthetists' ultrasound scanning for regional anaesthesia.

DETAILED DESCRIPTION:
This is a randomised, blinded interventional prospective study which will be conducted and reported as per the Consolidated Standards of Reporting Trials - Artificial Intelligence (CONSORT-AI) guidance. The study end points have been defined prospectively, and data will be divided into two cohorts (with vs without ScanNav Anatomy PNB assistance). Participants will be asked to perform ultrasound (US) scanning on healthy volunteers while under observation by a subject matter expert (expert observer) who will assess participant performance, both with and without the device. The US scans will be recorded and blinded expert observers (without knowledge of whether ScanNav Anatomy PNB is in use) will also assess acquisition of an appropriate block view (panel of three experts, one viewing each scan as per the unblinded assessors). The initial assessment will be undertaken after a scanning tutorial and then repeated after 8-10 weeks (to assess longer-term impact of the device).

ELIGIBILITY:
Inclusion Criteria:

1. Anaesthetist in Stage 1 of UK Anaesthesia Core/Specialty Training (CT 1-3)
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study
3. Available to travel and attend the study day in person

Exclusion Criteria:

1. Aged <18 years of age
2. Unwilling or unable to provide informed consent
3. Expert in UGRA (see definition above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 70 participants will be recruited to represent the intended user population (anaesthetists qualified to perform UGRA, but non-experts in the field of regional anaesthesia).
  Potential study participants will be identified by approaching professional anaesthesia/anaesthetics societies, networks (e.g., Wales Regional Anaesthesia Group - South).
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Block identification (long-term) | 8-10 weeks
  Identification of an appropriate block view by participant [blinded expert's opinion; Y/N] both with and without the use of ScanNav Anatomy PNB for ultrasound scanning (8 - 10 weeks after teaching)

SECONDARY OUTCOMES:
Block identification (immediate) | Time 0
  Identification of an appropriate block view by participant [blinded expert's opinion; Y/N] both with and without the use of ScanNav Anatomy PNB for ultrasound scanning (immediately after teaching)
Anatomy identification | Time 0 and 8-10 weeks
  Correct identification of anatomical structures on the block view [Y/N]
Participant confidence | Time 0 and 8-10 weeks
  Participant confidence in ultrasound scanning [continuous scale; 0 (no confidence] - 10 (total confidence)]
Overall scan performance | Time 0 and 8-10 weeks
  Expert observer's assessment of the participant's overall ultrasound scanning performance [continuous scale; 0 (poor) - 10 (excellent)]

CONTACTS AND LOCATIONS:
Overall Officials: James Bowness, Dr, Principal Investigator — Intelligent Ultrasound
Locations (1):
- UCH Education Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kowa CY, Morecroft M, Macfarlane AJR, Burckett-St Laurent D, Pawa A, West S, Margetts S, Haslam N, Ashken T, Sebastian MP, Thottungal A, Womack J, Noble JA, Higham H, Bowness JS. Prospective randomized evaluation of the sustained impact of assistive artificial intelligence on anesthetists' ultrasound scanning for regional anesthesia. BMJ Surg Interv Health Technol. 2024 Oct 16;6(1):e000264. doi: 10.1136/bmjsit-2024-000264. eCollection 2024. PMID 39430867